CLINICAL TRIAL: NCT00083759
Title: A Phase II, Multicenter, Double-blind, Placebo-Controlled Study of the Efficacy, Safety, and Tolerability of Intravenous Natalizumab (300 mg) in Subjects With Moderate to Severe Rheumatoid Arthritis (RA) Receiving Concomitant Treatment With Methotrexate (MTX)
Brief Title: Natalizumab in the Treatment of Rheumatoid Arthritis in Subjects Receiving Methotrexate
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The biological effect seen with natalizumab was not sufficient to warrant further development in RA.
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ELN100226-RA201
Record Dates: First submitted 2004-06-01; First posted 2004-06-03 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2009-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Natalizumab

ARMS (2):
- natalizumab (Active Comparator)
  Interventions: Drug: natalizumab
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: natalizumab
  Other Names: TYSABRI
  Arms: natalizumab
Drug: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability and efficacy of natalizumab in subjects diagnosed with moderate to severe rheumatoid arthritis (RA) receiving concomitant treatment with methotrexate (MTX). It is thought that natalizumab may stop the movement of certain white blood cells, known as lymphocytes, into joint tissue. These cells are thought to cause damage in the joints leading to the symptoms of RA.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible to begin study participation if they meet all of the following inclusion criteria:

* Subject is able to read, understand, and voluntarily sign the approved Informed Consent form prior to the performance of any study-specific procedures;
* Male or female subjects, ≥18 to ≤75 years of age, who has a diagnosis of rheumatoid arthritis Functional Class 1 to 3 by the 1987 Revised American Rheumatism Association Criteria for the Classification of Rheumatoid Arthritis for at least 6 months prior to screening;
* Subject is on a stable dose of MTX of at least 10 mg/week for ≥3 months prior to randomization (Month 0) without an adequate response;
* Female subjects of childbearing potential agree to use adequate, contraceptive methods (either intrauterine device [IUD], oral or depot contraceptive, or barrier plus spermicide). Female subjects of childbearing potential use adequate contraception for at least 2 months prior to study entry and continue contraception for at least 3 months after their last infusion of study drug;
* Subject is willing and able to complete all planned study procedures;
* Subject has at least 10 painful/tender and 6 swollen joints at the Month 0 (Baseline) visit;
* Subject has an elevated CRP level (defined as >2.87 mg/L) at Screening.

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the following exclusion criteria:

* Subject is pregnant or lactating;
* Subject who has experienced an inadequate therapeutic response after at least 3 months of treatment with at least one TNF-alpha inhibitor;
* Subject who has received treatment with anakinra;
* Subject who has received prior treatment with natalizumab;
* Subject does not meet the following criteria regarding concomitant medications for RA:
* Use of any oral steroid exceeding 10 mg/day of prednisone (or equivalent dose) and not administered at a stable dose for at least 1 month prior to randomization (Month 0);
* Use of any NSAIDs unless stable for at least 1 month prior to randomization (Month 0);
* Use of other anti-arthritic treatments, including approved or experimental oral, topical, or injectable biologics or drugs, or devices within 1 month prior to randomization (Month 0);
* Intra-articular corticosteroid injections within 1 month prior to randomization (Month 0);
* Treatment with any TNF-alpha inhibitor within 2 months prior to randomization (Month 0);
* Subject who is expected to be unavailable for the duration of the trial, likely to be noncompliant with the Protocol, or felt to be unsuitable by the Investigator for any other reason;
* Subject who has a history of a malignancy (other than basal cell carcinoma of the skin);
* Subject who has a history of clinically significant and/or persistent gastrointestinal, pulmonary, chronic infection, cardiovascular, renal, hepatic, neurological, dermatological, immunological, major psychiatric (including drug or alcohol abusers) or hematological illness, which, in the opinion of the Investigator placed the subject at unacceptable risk for participation in the study;
* Subject who has any laboratory test at Screening considered significantly abnormal. An alanine transaminase (ALT) or aspartate transaminase (AST) ≥1.5 x upper limits of normal (ULN) and cytopenia (included any of the following: WBC <3.5 x 1000/uL; hemoglobin [Hb] <8 g/dL; platelets <100 x 1000/uL; and/or neutrophils absolute <1.0 x 1000/uL) were considered significantly abnormal;
* Subject who intends to donate blood or blood products during the period of the study or within 1 month following completion of the study;
* Subject who has a positive tuberculosis (TB) skin test at Screening or within the 30 days prior to Screening (defined as ≥10 mm induration);
* Subject who plans or requires any surgical procedure during the study treatment period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2004-05; Primary Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Clinical Research Unit / University of Arizona, Tucson, Arizona
  - Arthritis Medical Clinic of North County, Inc., Escondido, California
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Massachusetts General Hospital, Boston, Maine
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Justus Fiechtner, MD, PC, Lansing, Michigan
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Rheumatic Disease Associates, Willow Grove, Pennsylvania
  - Radiant Research, Dallas, Texas
- Canada (2):
  - St. Clare's Mercy Hospital, St. John's, Newfoundland and Labrador
  - The Arthritis Program Research Group Inc., Newmarket, Ontario

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient entered 24 May 2004, study terminated 28 February 2005. A total of 299 patients were evaluable for safety and 273 patients for efficacy. Study conducted in Argentina, Australia, Canada, Czech Republic, Poland, Slovakia, and the United States.
Pre-assignment Details: Patients who met these criteria were randomized to natalizumab or placebo: aged 18-75 with a diagnosis of rheumatoid arthritis (RA) Functional Class 1-3 for ≥ 6 months, on a stable dose of methotrexate (MTX), having ≥ 10 painful/tender joints, and with elevated C-reactive protein. Stratification based on baseline number of painful/tender joints.
Groups:
- Natalizumab: Natalizumab 300 mg as monthly IV infusions + methotrexate (MTX)
- Placebo: Placebo IV infusions + methotrexate (MTX)
Period: Overall Study
Arm/Group | Natalizumab | Placebo
Started | 150 (150 subjects enrolled, 137 (Modified Intention-to-Treat [MITT] Population) for efficacy analyses) | 149 (149 subjects enrolled, 136 (Modified Intention-to-Treat [MITT] Population) for efficacy analyses)
Completed | 66 | 66
Not Completed | 84 | 83
Not completed — Adverse Event | 5 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 1 | 1
Not completed — Inadequate Therapeutic Response | 32 | 35
Not completed — Subject Withdrew Consent | 2 | 2
Not completed — Non-Compliance | 1 | 0
Not completed — Sponsor's Discretion | 28 | 29
Not completed — Other | 14 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Natalizumab | Placebo | Total
Number analyzed (Participants) | 137 | 136 | 273
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (10.5) | 53.6 (10.4) | 52.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 107 | 218
  Male | 26 | 29 | 55
Baseline Count of Painful/Tender Joints [Number; unit: participants]
  <20 | 44 | 43 | 87
  >20 | 93 | 93 | 186

OUTCOME MEASURES:

1. Primary Outcome: American College of Rheumatology (ACR)20.
Description: ≥20% reduction from baseline in painful/tender joint count and swollen joint count and ≥20% improvement in at least three of five secondary clinical parameters (e.g., subject global assessment, physician global assessment, pain scale, disability score, and an acute phase reactant)
Time Frame: Month 6
Measure: Number; unit: participants
Arm/Group | Natalizumab | Placebo
Number analyzed (Participants) | 137 | 136
participants | 59 | 45
Statistical Analysis 1: Comparison: Natalizumab vs Placebo; Test type: Superiority or Other; p = 0.089, Cochran-Mantel-Haenszel

2. Secondary Outcome: American College of Rheumatology (ACR)50
Description: ≥50% reduction from baseline in painful/tender joint count and swollen joint count and ≥50% improvement in at least three of five secondary clinical parameters (e.g., subject global assessment, physician global assessment, pain scale, disability score, and an acute phase reactant)
Time Frame: Month 6
Measure: Number; unit: participants
Arm/Group | Natalizumab | Placebo
Number analyzed (Participants) | 137 | 136
participants | 23 | 15
Statistical Analysis 1: Comparison: Natalizumab vs Placebo; Test type: Superiority or Other; p = 0.171, Cochran-Mantel-Haenszel

3. Secondary Outcome: American College of Rheumatology (ACR)70
Description: ≥70% reduction from baseline in painful/tender joint count and swollen joint count and ≥70% improvement in at least three of five secondary clinical parameters (e.g., subject global assessment, physician global assessment, pain scale, disability score, and an acute phase reactant)
Time Frame: Month 6
Measure: Number; unit: participants
Arm/Group | Natalizumab | Placebo
Number analyzed (Participants) | 137 | 136
participants | 13 | 10
Statistical Analysis 1: Comparison: Natalizumab vs Placebo; Test type: Superiority or Other; p = 0.526, Cochran-Mantel-Haenszel

LIMITATIONS AND CAVEATS:
The study was terminated prematurely on 28 February 2005. The biological effect seen with natalizumab was not sufficient to warrant further development in RA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor will have at least 30 days to request revisions to a proposed Publication. Institution will delete any Confidential Information provided by Sponsor, will delay Publication submission for a further 90 days for the filing of patent applications, and will not issue a press release about the Study without the Sponsor's prior written consent.